CLINICAL TRIAL: NCT04577196
Title: Impact of Information Processing Via a Dashboard on the Situational Awareness of the Trauma Team Prior to the Management of a Critical Patient: an Experimental Simulation Study
Brief Title: Improving Situational Awareness Before Acute Care
Acronym: IMPULSE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC
Record Dates: First submitted 2020-09-25; First posted 2020-10-06 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Critical Illness; Trauma
Keywords: Simulation training; Non-technical skills; Data processing; Trauma team briefing; Situational awareness; Cognitive support
MeSH Terms: conditions — Critical Illness; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Briefing supported by the trauma dashboard: During the entire chain of transmission (from the initial phone call to the end of the briefing to the trauma team) the trauma leader will be provided with a trauma dashboard to synthesize and disseminate the available information about the arriving patient.
  Interventions: Other: Trauma dashboard
- Briefing without the trauma dashboard: The transmission chain will not be supported by any specific tool.

INTERVENTIONS:
Other: Trauma dashboard — A large dashboard available to all, providing a framework for synthesizing and displaying relevant information about the arriving critical patient, to be filled in by the trauma leader.
  Groups: Briefing supported by the trauma dashboard

SUMMARY:
This study aims to assess the impact on the trauma team's situational awareness of using a dashboard to synthesize and disseminate available information on a critical patient incoming to the trauma center.

DETAILED DESCRIPTION:
This trial will be carried out at the Grenoble Alpes University Hospital's simulation center. Volunteer professionals will run scenarios simulating the information transmission chain "pre-hospital team - trauma leader - trauma team" just prior to the admission of a critical patient to the trauma center. In each scenario, the trauma leader will be alerted by phone that a patient is being managed by a pre-hospital medical team and is about to be transferred to the trauma center. The trauma leader will have to synthesize and disseminate the available information to the trauma team (composed of a junior physician, a resident and a nurse). Depending on the allocation group, the transmission chain will be supported or not by a specific trauma dashboard. The scenario will be discontinued at the end of this handover and before the patient's arrival.

ELIGIBILITY:
Inclusion Criteria:

* Physicians, residents and nurses from the Grenoble Alpes University Hospital volunteering to participate.

Exclusion Criteria:

* Prior knowledge of the study scenarios
* Study investigator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physicians, residents and nurses from the Grenoble Alpes University Hospital volunteering to participate.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Trauma team situational awareness | immediately after the end of the information transmission
  Situational Awareness Global Assessment Technique questionnaire (score from 0 to 15/15, higher scores mean a better situational awareness)